CLINICAL TRIAL: NCT05540626
Title: Real World Evidence Study Utilizing the Cala Trio Device in Patients With Essential Tremor
Brief Title: RWE Study Utilizing the Cala Trio Device in Patients With Essential Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cala Health, Inc. (Industry)
Collaborators: CVS Healthspire Life Sciences Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Aetna RWE
Record Dates: First submitted 2022-09-02; First posted 2022-09-14 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care Arm (No Intervention): Baseline tremor power without stimulation (SOC arm) over the first month of the study. Subjects in the SOC arm will be asked to measure their tremor severity by doing daily postural holds with the Cala Trio device without actual stimulation.
- Intervention with the Cala Trio device (CTD) arm (Experimental): Tremor power after stimulation with Cala Trio. Subjects in the intervention arm will wear the device at home for a period of 12 months, during which they will deliver 40 min stimulation sessions, which can be started and stopped on demand.
  Interventions: Device: Cala Trio

INTERVENTIONS:
Device: Cala Trio — transcutaneous afferent patterned stimulation (TAPS)
  Arms: Intervention with the Cala Trio device (CTD) arm

SUMMARY:
The study objective is to evaluate hand tremor relief in the treated hand following stimulation with the Cala Trio Device in adults with essential tremor, and healthcare resource utilization and total healthcare costs over a 12-month period.

DETAILED DESCRIPTION:
This is a prospective, randomized, dual arm, pragmatic trial in a real-world setting to evaluate the effectiveness and health economics outcomes of the Cala Trio device in reducing hand tremor and improving quality of life as measured by the Bain and Findley Activities of Daily Living (ADL) score relevant to the stimulated upper limb. Healthcare resources utilization and total all-cause healthcare will also be evaluated. The study will recruit approximately 300 patients: 150 in the intervention arm (Cala Trio device)and 150 patients in the standard of care (SOC) arm. Subjects will be randomized to either the intervention arm or the standard of care arm (1:1).Subjects in the SOC arm will be asked to measure their tremor severity by doing daily postural holds with the Cala Trio device without actual stimulation. Subjects in the intervention arm will wear the device at home for a period of 12 months, during which they will deliver 40 min stimulation sessions, which can be started and stopped on demand. After the first month, the subjects who were randomized to the SOC arm will cross over to the intervention arm.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥22years
* Aetna commercial fully insured OR Medicare Advantage population (inclusion of Medicare is contingent upon additional internal approvals)
* Two ICD claims for ET, at least seven days apart, in the last three years OR one ICD claim for ET followed by at least one dispensed pharmaceutical treatment for ET
* Contraindication to standard pharmacological therapy (Asthma, COPD, 1stor 2nddegree heart block) OR indicator of poor pharmacological acceptability as evidenced by drug switching behaviors OR indicator of drug resistance as evidenced by the use of third-line drug therapies including Clozapine, Mirtazapine, Gabapentin, Topiramate, Clonazepam or Alprazolam
* Willing and able to provide informed consent to participate in the study
* Willing and able to follow study protocol requirements
* Patients with PCP or neurologist provider encounter in past 18months

Exclusion Criteria:

* ICD-10 evidence of a pacemaker or defibrillator or a procedure code indicating pacemaker implantation, electrode renewal or calibration
* ICD-10 evidence of a deep brain stimulator or a procedure code indicating DBS implantation
* CPT/HCPCS evidence of thalamotomy, gamma-knife radio surgical thalamotomy
* NDC and CPT evidence of botulinum toxin the last 6 months as therapeutic injection in the upper limb
* Pregnant during the enrollment period
* Evidence of Parkinson's Disease
* Evidence of epilepsy
* Formal diagnosis of hypothyroidism and treatment
* Formal diagnosis of hyperthyroidism without evidence of treatment
* Formal diagnosis of dementia
* Evidence of Treatment with thyroid hormone supplements (2 Rx claims 28 or more days apart) or evidence of hyperthyroidism (2+ claims, 28 days or more apart)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change in tremor power | 1 Month
  Difference in tremor power after stimulation with Cala Trio (treated arm) and baseline tremor power without stimulation (SOC arm) over the first month of the study.
  Prior to and immediately after each of the first 40 stimulation sessions and every 7th session thereafter, the Cala Trio will direct the patient to perform postural hold tremor tasks to measure tremor power pre and post stimulation. The SOC arm will perform a tremor measurement only, without any stimulation sessions, for 1 month.

SECONDARY OUTCOMES:
Bain & Findley Activities of Daily Living (BF-ADL) scale subset score | 12 Months
  BF-ADL subset score relevant to the stimulated upper limb. The subset score is the sum of 8 rated tasks. Each task is rated 1 to 4, where a higher score indicates more severe tremor. Minimum subset score = 8; Maximum subset score = 32. Improvements in BF-ADL scores will be measured from baseline over the 12 months study duration.
Tremor power improvement ratio (TPIR) | 12 Months
  TPIR is defined as the ratio of pre- to post-stimulation tremor power. Per-patient median TPIR over first, second, third, and fourth quarters of the study (i.e., months 1 - 3, 4 - 6, etc.) will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Cala Health, San Mateo, California, United States

REFERENCES:
- [Derived] Brillman S, Khemani P, Isaacson SH, Pahwa R, Deshpande R, Zraick V, Rajagopal A, Khosla D, Rosenbluth KH. Non-Invasive Transcutaneous Afferent Patterned Stimulation Therapy Offers Action Tremor Relief in Parkinson's Disease. Tremor Other Hyperkinet Mov (N Y). 2023 Aug 23;13:25. doi: 10.5334/tohm.762. eCollection 2023. PMID 37637850